CLINICAL TRIAL: NCT00712075
Title: Functional Rehabilitation for Older Patients With Schizophrenia (FROPS)
Brief Title: Functional Rehabilitation for Older Patients With Schizophrenia
Acronym: FROPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E4876-R
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia; Aging
Keywords: Cognitive Behavioral Therapy; Social Skills Training; Experience Sampling Method; Computer-assisted therapy; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBSST+PDA (Experimental): PDA-Assisted Cognitive-Behavioral Social Skills Training (CBSST+PDA): The CBSST rehabilitation intervention will be combined with the use of a PDA to facilitate homework completion and progress towards recovery goal attainment in consumers.
  Interventions: Behavioral: CBSST+PDA
- CBSST (Active Comparator): Cognitive Behavioral Social Skills Training (CBSST): CBSST is a psychosocial rehabilitation intervention that combines skills from cognitive behavioral therapy and social skills training to assist consumers in improving functioning and recovery goal attainment.
  Interventions: Behavioral: Cognitive Behavioral Social Skills Training
- PDA-Only (Active Comparator): PDA-only: To control of device contact, the PDA-only arm will not receive CBSST and will only carry a PDA with access to the basic features of the device.
  Interventions: Behavioral: PDA-only

INTERVENTIONS:
Behavioral: CBSST+PDA — PDA-Assisted Cognitive Behavioral Social Skills Training (CBSST+PDA) includes weekly group therapy sessions, each 90 minutes in length, with 6-8 patients (maximum of 10) were held for 24 weeks. The intervention integrated cognitive behavioral and social skills training interventions modified for use with older patients with psychosis. Participants utilized PDAs to assist with homework completion and compliance.
  Other Names: PDA-Assisted Cognitive Behavioral Social Skills Training
  Arms: CBSST+PDA
Behavioral: Cognitive Behavioral Social Skills Training — Cognitive Behavioral Social Skills Training includes weekly group therapy sessions, each 2.5 hours (30 min lunch break) in length, with 6-8 patients (maximum of 10) were held for 24 weeks. The intervention integrated cognitive behavioral and social skills training interventions modified for use with older patients with psychosis.
  Other Names: CBSST
  Arms: CBSST
Behavioral: PDA-only — To control for the effects of having a PDA, a third group was provided PDAs for the same duration as the other two groups. Participants had access to the same basic functions (calendar, contact list, etc.) as the CBSST+PDA group, but did not have any homework or weekly group meetings.
  Arms: PDA-Only

SUMMARY:
Aging and psychosis are major priority areas for VA. This project is a continuation of a Merit Review Program, in which we developed, manualized and conducted randomized controlled trials of a novel psychosocial rehabilitation intervention for older people with schizophrenia, called cognitive-behavioral social skills training (CBSST). We found that CBSST improved community functioning in these patients. CBSST, however, is an intensive program that would burden VA mental health clinics with demands for additional staff and financial resources and burdens older veterans with travel and time demands. To reduce these burdens and barriers to implementation of CBSST, we are developing a computer-assisted CBSST intervention that takes advantage of available handheld computer technology. Therapist contact is cut 50% and replaced by handheld computer-assisted CBSST intervention tools. The project will examine whether computer-assisted CBSST is as effective as the full CBSST program, while improving client satisfaction and reducing burden and cost.

DETAILED DESCRIPTION:
Aging and psychosis are major priority areas for VA. This project is a continuation of a Merit Review Program, in which we developed, manualized and conducted randomized controlled trials of a novel psychosocial rehabilitation intervention for older people with schizophrenia, called cognitive-behavioral social skills training (CBSST). We found that CBSST improved community functioning in these patients. CBSST, however, is an intensive program that may burden VA mental health clinics with demands for additional staff and financial resources and Veterans with travel and time demands. To reduce these burdens and barriers to implementation of CBSST, we developed a computer-assisted CBSST intervention that takes advantage of available handheld computer technology (personal data assistants or PDAs). Therapist contact is cut 50% and replaced by handheld computer-assisted CBSST intervention tools. The project will examine whether computer-assisted CBSST is as effective as the full CBSST program, while improving client satisfaction and reducing burden and cost. A randomized-controlled clinical trial comparing 3 treatment conditions (computer-assisted CBSST, CBSST, and a PDA-only control condition) will be conducted. Participants will be recruited, treated for 6 months and followed longitudinally for 6 months after treatment. A multidimensional evaluation of treatment outcome, including functioning (primary outcome), CBSST skills acquisition, and symptoms will be conducted at baseline, mid-treatment, end of treatment (6-months after baseline), and 6-month follow-up (12 months after baseline). Factors that might mediate improvement in CBSST will be assessed, including homework adherence, cognitive insight (metacognition and belief flexibility), and defeatist performance beliefs (e.g., "Why try, I'll just fail again").

The proposed project will also use innovative computer-assisted Ecological Momentary Assessment (EMAc) methods to measure outcomes. EMAc is an ambulatory data collection technique that permits the real time, real world monitoring of behaviors, moods, and cognitions. Participants are signaled by handheld computers several times throughout the day to respond to questionnaires, which eliminates recall and information-processing biases that can compromise the validity of traditional self-report and interview measures. Outcomes in the proposed trial will be assessed using traditional measures, as well as EMAc measures.

Specific Aims: (1) To determine whether computer-assisted CBSST is as effective as the full CBSST program (in prior project) and supportive contact, despite reduced burden and cost. (2) To examine whether EMAc measures of functioning and psychotic symptoms are sensitive to change in CBSST. (3) To examine whether increased cognitive insight, reduced defeatist performance beliefs, and greater homework adherence mediate outcomes in CBSST.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or Schizoaffective Disorder and age >45 (Veterans and non-Veterans)
* fluency in English
* Medical, psychiatric and substance abuse sufficiently stable for outpatient group therapy

Exclusion Criteria:

* prior exposure to CBST during the previous 5 years

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Granholm, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included 77 community dwelling Veterans and non-Veterans. Inclusion criteria: diagnosis of schizophrenia or schizoaffective, age 45 or older, fluency in English, and medical, psychiatric and substance abuse sufficiently stable for outpatient group therapy Exclusion criteria: prior exposure to CBT during the previous five years.
Pre-assignment Details: 107 participants were enrolled in the study and 77 participants started the study. 30 were excluded (lost interest, N=6; Wrong diagnosis, N=10; Early study termination, N=4; Medically unstable, N=2; Psychiatrically unstable, N=4; Prior CBT, N=4).
Period: Overall Study
Arm/Group | CBSST+PDA | CBSST | PDA-Only
Started | 22 | 30 | 25
Completed | 17 | 26 | 14
Not Completed | 5 | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBSST+PDA | CBSST | PDA-Only | Total
Number analyzed (Participants) | 17 | 26 | 14 | 57
Age, Customized [Number; unit: participants]
  Age 45 and older | 17 | 26 | 14 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 1 | 10
  Male | 16 | 18 | 13 | 47
Region of Enrollment [Number; unit: participants]
  United States | 17 | 26 | 14 | 57

OUTCOME MEASURES:

1. Primary Outcome: Independent Living Skills Survey (ILSS)
Description: The ILSS is a self-report measure in an interview format to assess everyday functioning in ten domains: Appearance and Clothing, Personal Hygiene, Care of Personal Possessions, Food Preparation/Storage, Health Maintenance, Money Management, Transportation, Leisure, Job Seeking, and Job Maintenance. Scale ranges from 0 to 1. Subscales are averaged to yield composite score. Higher scores represent a higher level of functioning.
Time Frame: Baseline, at mid-treatment (3-mo), at end-of-treatment (6-mos), and at 6-mo follow-up (12 mos post-baseline)
Population: Due to incomplete ILSS data for one participant in the CBSST group, 25 of 26 participants were included in the analyses for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST+PDA | CBSST | PDA-Only
Number analyzed (Participants) | 17 | 25 | 14
units on a scale
  Baseline | 0.69 (0.10) | 0.67 (0.09) | 0.71 (0.10)
  3 months | 0.69 (0.10) | 0.69 (0.09) | 0.73 (0.10)
  6 months | 0.71 (0.10) | 0.70 (0.09) | 0.69 (0.12)
  12 months | 0.67 (0.14) | 0.71 (0.9) | 0.70 (0.13)

2. Secondary Outcome: Comprehensive Module Test (CMT)
Description: The Comprehensive Module Test (CMT) is an assessment of CBSST skills acquisition in three domains: Communication Skills Test, Problem Solving Test, and Thought Challenging Test. The total CMT score ranges from 0-33. Higher total scores represent higher level of CBSST skills acquisition.
Time Frame: Baseline, at mid-treatment (3-mo), at end-of-treatment (6-mos), and at 6-mo follow-up (12 mos post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST+PDA | CBSST | PDA-Only
Number analyzed (Participants) | 17 | 26 | 14
units on a scale
  Baseline | 4.3 (3.6) | 5.8 (2.9) | 3.9 (3.5)
  3 months | 4.3 (3.6) | 5.8 (2.9) | 3.9 (3.5)
  6 months | 8.4 (5.7) | 11.0 (5.3) | 3.3 (2.3)
  12 months | 4.3 (2.7) | 9.1 (5.8) | 1.7 (2.1)

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The PANSS is 30 item semi-structured clinical interview designed to assess positive and negative symptoms. The PANSS consists of 7 items on the positive symptom subscale, 7 items on the negative symptom subscale, and 16 items on the general psychopathology subscale. Each item in the subscale is rated from 0 (absence of symptom) to 7 (extreme symptom severity). Scores of each subscale are summed to yield a total score range of 30 (Absence of symptoms) to 210, where higher scores represent more severe symptoms.
Time Frame: Baseline, at mid-treatment (3-mo), at end-of-treatment (6-mos), and at 6-mo follow-up (12 mos post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST+PDA | CBSST | PDA-Only
Number analyzed (Participants) | 17 | 26 | 14
units on a scale
  Baseline | 68.6 (22.3) | 72.0 (25.4) | 70.6 (20.9)
  3 months | 66.8 (19.4) | 65.3 (24.9) | 58.2 (17.9)
  6 months | 62.2 (18.5) | 61.0 (17.8) | 62.9 (17.3)
  12 months | 63.5 (19.9) | 61.8 (21.4) | 68.0 (13.7)

ADVERSE EVENTS:
Arm/Group | CBSST+PDA | CBSST | PDA-Only
Serious Adverse Events (participants affected / at risk) | 0/22 | 4/30 | 0/25
Other Adverse Events (participants affected / at risk) | 0/22 | 0/30 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBSST+PDA (N=22) | CBSST (N=30) | PDA-Only (N=25)
Hospitalization (Psychiatric disorders) | 0 | 4 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small sample size and loss of follow-up data.

No 50% CBSST comparison group without mobile computer to test efficacy of shorter treatment alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes